CLINICAL TRIAL: NCT00071396
Title: Continuous Infusion Followed by Subcutaneous Injection of Campath-1H Plus Rituximab in the Treatment of CD52- and CD20-Positive Refractory or Relapsed Chronic Lymphoid Disorders
Brief Title: Campath-1H Plus Rituximab for CD52- and CD20- Positive Refractory or Relapsed Chronic Lymphoid Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-368
Record Dates: First submitted 2003-10-21; First posted 2003-10-22 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CD-52 and CD-20 Positive; Refractory; Relapsed
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — Alemtuzumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Campath-1H + Rituximab (Experimental): Campath 15 mg/day continuous intravenous (IV) infusion x 6 days, then twice a week for 3 weeks as 30 mg injection under skin to complete 4 week treatment course.
  Rituximab 375 mg/m^2 IV infusion day 1, then 500 mg/m^2 on days 8, 15 + 22.
  Interventions: Drug: Campath-1H; Drug: Rituximab

INTERVENTIONS:
Drug: Campath-1H — 15 mg/day Continuous infusion by vein (IV) for 6 days then given twice a week for remaining three weeks as 30 mg injection under skin to complete one treatment course of 4 weeks.
  Other Names: Alemtuzumab; Campath
Drug: Rituximab — 375 mg/m^2 IV infusion on day 1, then 500 mg/m^2 on days 8, 15, and 22.
  Other Names: Rituxan

SUMMARY:
The goal of this clinical research study is to learn if giving CAMPATH-1H with rituximab can shrink or slow the growth of the disease in patients with chronic lymphoid disorders that have either not responded or whose disease has returned after treatment with standard therapies.

DETAILED DESCRIPTION:
Objectives:

1. To determine the efficacy and response rates of Campath-1H when given as a continuous intravenous infusion followed by subcutaneous injection plus rituximab in the treatment of chronic lymphoid disorders that are refractory to conventional therapy, have relapsed, or have no established frontline therapy.
2. To assess the safety of the combination of Campath-1H when given as a continuous intravenous infusion followed by subcutaneous injection plus rituximab in chronic lymphoid disorders that express both CD52 and CD20 cell surface antigens.
3. To measure levels of soluble (s) CD20 and sCD52 as well as levels of Campath-1H, rituximab and antibody complexes of rituximab/CD20 and Campath-1H/CD52 in patients with chronic lymphoid disorders treated with Campath-1H plus rituximab.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/=15 years.
2. Written informed consent.
3. Patients with chronic lymphoid malignancies that are either refractory to frontline therapy or have relapsed and that have a predicted probability of response of less than 20% with conventional therapy or allogeneic/autologous stem cell transplantation.
4. The following histologies are included: B-cell chronic lymphocytic leukemia (B-CLL or B-cell CLL), B-cell prolymphocytic leukemia (PLL), chronic lymphoid leukemia (CLL/PLL), hairy cell leukemia and hairy cell variant, mantle cell leukemia/lymphoma, marginal zone lymphoma/leukemia, splenic lymphoma with villous lymphocytes, CLL with evidence of transformation (e.g., Richter's transformation), large granular lymphocytic leukemia (LGL and NK-cell type).
5. Patients with above mentioned histologies whose malignant cell population have expressed both CD52 and CD20 in >/= 20% of cells as assessed by flow cytometry or immunohistochemistry. Expression of CD20 or CD52 < 20% is permitted if patients received rituximab or alemtuzumab, respectively, within 3 months prior to study start.

Exclusion Criteria:

1. Patients who have previously received Rituximab and CAMPATH-1H in combination are excluded.
2. ECOG performance status of </= 2.
3. Serum creatinine </= 2mg/dL and total bilirubin of £ 2 mg/dL unless due to direct infiltration of the liver or kidney with malignant cells.
4. Patients with a past history of anaphylaxis following exposure to rat or mouse derived CDR-grafted humanized monoclonal antibodies are excluded <CDR = complementarity determining regions>.
5. Negative pregnancy test (serum or urine) if female and of childbearing potential only (non-childbearing is defined as greater than one year post-menopausal or surgically sterilized).
6. No prior chemotherapy, immunotherapy, or hormonal therapy within 2 weeks prior to study start. Hormonal replacement therapy is permitted. No prior therapy with monoclonal antibodies for at least 4 weeks prior to study start.
7. Patients at high risk of hepatitis B virus (HBV) infection and active HBV infection are excluded.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-10; Primary Completion 2006-09 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center's website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 10/21/02 - 3/27/09; all patients were registered at the University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of 48 patients enrolled, 41 patients were evaluable for response (2 patients withdrew before starting treatment and 2 were ineligible).
Groups:
- Campath-1H + Rituximab: Campath 15 mg/day continuous intravenous (IV) infusion for 6 days, then twice a week for 3 weeks as 30 mg injection under skin to complete 4 week treatment course.
  Rituximab 375 mg/m^2 IV infusion day 1, then 500 mg/m^2 on days 8, 15 + 22.
Period: Overall Study
Arm/Group | Campath-1H + Rituximab
Started | 44
Completed | 41 (Evaluable for response.)
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Campath-1H + Rituximab
Number analyzed (Participants) | 44
Age Continuous [Median (Full Range); unit: years] | 59 [39 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Overall response categorized as 'Complete Remission,' 'Partial Remission,' or 'No Response.' Blood tests weekly while on active therapy, within 4-6 weeks following last dose of therapy, and every 3 to 6 (+/- month) thereafter as long as on study. Repeat bone marrow biopsy/aspirate with flow cytometry as applicable at the end of first course of therapy, (1 week) within 4-6 weeks following the last dose of therapy and every 6 to 12 months (+/-) thereafter as long as on study.
Time Frame: After each 4 week course of treatment
Population: Analysis treated population 41 evaluable patients (44 treated, 3 not evaluable for response).
Measure: Number; unit: Participants
Arm/Group | Campath-1H + Rituximab
Number analyzed (Participants) | 41
Participants
  Complete Remission | 8
  Partial Remission | 14
  No Response | 19

ADVERSE EVENTS:
Time Frame: 3 years 11 months
Arm/Group | Campath-1H + Rituximab
Serious Adverse Events (participants affected / at risk) | 8/44
Other Adverse Events (participants affected / at risk) | 25/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Campath-1H + Rituximab (N=44)
Fever without neutropenia (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 3 (3)
Febrile Neutropenia (Infections and infestations) | 3 (3)
Fever (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Campath-1H + Rituximab (N=44)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Drug Fever (General disorders) | 12 (13)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
fatigue (General disorders) | 10 (10)
febrile neutropenia (General disorders) | 3 (3)
fever (General disorders) | 3 (5)
hypotension (Cardiac disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 8 (8)
puritis (Skin and subcutaneous tissue disorders) | 7 (7)
Injection site reaction (Skin and subcutaneous tissue disorders) | 5 (8)
Leukopenia (Blood and lymphatic system disorders) | 9 (12)
Lymphopenia (Blood and lymphatic system disorders) | 7 (7)
neutropenia (Infections and infestations) | 3 (5)
Rigors Chills (General disorders) | 18 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No